CLINICAL TRIAL: NCT02220296
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0123-0338 in Healthy Subjects and in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1438-4137; 2014-000071-70 (EudraCT Number); U1111-1151-9327 (Other: WHO)
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Healthy; Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 insulin 338 (Experimental)
  Interventions: Drug: Insulin 338
- Part 1 placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Part 2 insulin 338 (Experimental)
  Interventions: Drug: Insulin 338
- Part 2 insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: Insulin 338 — Healthy subjects will receive a single dose of insulin 338 in ascending doses. Injected subcutaneously (under the skin).
  Arms: Part 1 insulin 338
Drug: placebo — Healthy subjects will receive a single dose of placebo. Injected subcutaneously (under the skin).
  Arms: Part 1 placebo
Drug: Insulin 338 — Subjects with type 1 DM will receive a single dose of insulin 338 in ascending doses. Injected subcutaneously (under the skin).
  Arms: Part 2 insulin 338
Drug: insulin glargine — Subjects with type 1 DM will receive 0.4 U/kg insulin glargine once daily for 4 days. Injected subcutaneously (under the skin).
  Arms: Part 2 insulin glargine

SUMMARY:
This trial is conducted in Europe. The purpose is to evaluate safety and tolerability of a range of single doses of subcutaneous insulin 338.

ELIGIBILITY:
Inclusion Criteria:

* Trial Part 1 (Healthy subjects):
* Male subject
* Age 18-55 (both inclusive) at the time of signing inform consent
* Body mass index 19.0-29.9 kg/m^2 (both inclusive)
* Trial Part 2 (Subjects with type 1 diabetes mellitus):
* Male subject or female subject of non-child bearing potential. Non-child bearing potential: being surgically sterilized (i.e. tubal ligation, bilateral oopherectomies or hysterectomised) for more than 3 months or being postmenopausal (as defined by amenorrhoea for at least 2 years prior to screening and documented by follicle-stimulating hormone (FSH) 40 U/L)
* Age 18-64 years (both inclusive) at the time of signing inform consent
* Body mass index 19.0-29.9 kg/m^2 (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) for 12 months or longer
* Treated with multiple daily insulin injections or insulin pump treatment for 12 months or longer
* Glycated hemoglobin (HbA1c) 9.0% or less
* Fasting C-peptide less than 0.3 nmol/L

Exclusion Criteria:

* Trial Part 1 (healthy subjects):
* History of, or presence of, cancer, diabetes mellitus or any clinically significant cardiovascular, respiratory, metabolic (including dyslipidemia), renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Increased risk of thrombosis, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the investigator
* Currently smoke more than 1 cigarette per day (or the equivalent for other tobacco products) or smoking 1 cigarette or less per day and not considering being able to refrain from smoking or refrain from use of other types of nicotine products (e.g. such as chewing tobacco, nicotine gums) during the in-house periods
* Trial Part 2 (subjects with type 1 diabetes mellitus):
* History of, or presence of, cancer or any clinically significant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception of conditions associated with diabetes mellitus), haematological, dermatological, venereal, neurological, psychiatric, other major disorders or personal and/or family history of thromboembolism, as judged by the investigator
* Increased risk of thrombosis, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the investigator
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the past 6 months before start of this trial (screening)
* Cardiac problems defined as: 1) decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time, or 2) acute myocardial infarction at any time, or 3) angina pectoris within the last 12 months before start of this trial (screening)
* Currently smoke more than 1 cigarette per day (or the equivalent for other tobacco products) or smoking 1 cigarette or less per day and not considering being able to refrain from smoking or refrain from use of other types of nicotine products (e.g. such as chewing tobacco, nicotine gums) during the in-house periods.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day 1 - day 22

SECONDARY OUTCOMES:
Incidence of hypoglycaemic episodes | Day 1 - day 22
Area under the serum insulin 338 concentration-time curve from zero to infinity | Day 1- day 22
Maximum serum insulin 338 concentration observed | Day 1- day 22
Time for maximum serum insulin 338 concentration | Day 1- day 22
t1/2, the terminal half-life of insulin 338 | Day 1- day 22

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com